CLINICAL TRIAL: NCT02314481
Title: Deciphering Antitumour Response and Resistance With INtratumour Heterogeneity - DARWINII
Brief Title: Deciphering Antitumour Response and Resistance With INtratumour Heterogeneity
Acronym: DARWINII
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University College, London (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14/0274
Record Dates: First submitted 2014-12-05; First posted 2014-12-11 (Estimated); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Non-small Cell Lung Cancer
Keywords: NSCLC; Clonal dominance; Clonal evolution; Intratumour heterogeneity; Genomic instability; Drug resistance; Immunotherapy; PDL1; BRAF V600; ALK; RET; HER2 amplification; MPDL3280A; Vemurafenib; Alectinib; T-DM1; Trastuzumab emtansine; TRACERX
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Genomic Instability | interventions — atezolizumab; Vemurafenib; alectinib; Ado-Trastuzumab Emtansine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- No actionable mutation - MPDL3280A (Experimental): MPDL3280A 1200mg IV infusion - 3 weekly until progression or unacceptable toxicity.
  Or in combination with chemotherapy:
  * For non-squamous: Cisplatin or Carboplatin plus pemetrexed & MPDL3280A - 3 weekly for 4 cycles followed by MPDL3280A and pemetrexed 3 weekly until progression or unacceptable toxicity or completion of a total of 35 cycles. MPDL3280A will then continue 3 weekly until progression or unacceptable toxicity.
  * For squamous: Carboplatin plus paclitaxel & MPDL3280A - 3 weekly for 4 cycles followed by MPDL3280A 3 weekly until progression or unacceptable toxicity.
- BRAF V600 - vemurafenib (Experimental): Vemurafenib 960mg twice daily until PD
  Interventions: Drug: Vemurafenib
- ALK/RET gene rearrangement - alectinib (Experimental): Alectinib 600mg twice daily until PD
  Interventions: Drug: Alectinib
- HER2 amplification - T-DM1 (Experimental): Trastuzumab emtansine (T-DM1) 3.6mg/kg - 3 weekly until PD IV infusion
  Interventions: Drug: Trastuzumab emtansine

INTERVENTIONS:
Drug: MPDL3280A — Intravenous (IV) infusion, as monotherapy of in combination with chemotherapy
  Other Names: Atezolizumab
Drug: Vemurafenib — Film coated tablet
  Other Names: Zelboraf
  Arms: BRAF V600 - vemurafenib
Drug: Alectinib — capsule
  Other Names: Alecensa
  Arms: ALK/RET gene rearrangement - alectinib
Drug: Trastuzumab emtansine — Powder for concentrate for solution for infusion
  Other Names: T-DM1; Kadcyla
  Arms: HER2 amplification - T-DM1

SUMMARY:
DARWIN II is a multi-arm non-randomised phase II trial, Eligible patient will be those who relapse with NSCLC (clinical trials.gov ref. NCT02183883). .

The trial will investigate assess if intra-tumour heterogeneity (clonal vs subclonal actionable mutation) is associated with PFS.

Patients without an actionable mutation will receive MPDL3280A (atezolizumab), a monoclonal antibody targeting anti-PDL1, as monotherapy or in combination with chemotherapy, The options for combination therapy will vary depending on the histology of the NSCLC (i.e. non-squamous or squamous).

Patients with BRAFV600 mutations, HER2 Amplification, ALK/RET gene rearrangements will be enrolled into arms treating with vemurafenib, trastuzumab emtansine and alectinib respectively.

DARWIN II will include extensive exploratory biomarker analysis to investigate a number of genomic and immune markers that may predict response to MPDL3280A (atezolizumab) and help guide future clinical trial design.

DETAILED DESCRIPTION:
DARWIN II is an exploratory phase II study examining the role of intra-tumour heterogeneity and predicted neo-antigens on the anti-tumour activity of anti-PDL1 immunotherapy.

It will examine how clonal dominance and intratumour heterogeneity influence outcomes after treatment, offering a unique opportunity to decipher mechanisms of resistance to immunotherapy with anti-PDL1. These data will help improve future study design by developing greater understanding of patient selection for immunotherapies in patients with NSCLC. The relationship between intratumour heterogeneity and cfDNA/CTCs will also be explored in DARWIN II, which may develop tools for patient selection and monitoring to be examined further in future studies. Results from DARWIN II will help to identify a biomarker for anti-PD-L1 therapy which could be used for patient stratification in future phase III trials of molecules targeting this T-cell inhibitory checkpoint. DARWIN II will also provide preliminary data on efficacy of MPDL3280A, which could be used to design randomised studies.

This is a multicentre non-randomised phase II study based on patients with relapsed NSCLC, who have provided a biopsy sample at the time of relapse.

The study arms:

* Arm 1: Patients without an actionable mutation - MPDL3280A (atezolizumab) monotherapy or in combination with chemptherapy
* Arm 2: BRAFV600 - vemurafenib
* Arm 3: ALK/RET gene rearrangement - alectinib
* Arm 4: HER2 Amplification - trastuzumab emtansine

Arms 2-4 are closed to further recruitment as of 25th May 2021.

ELIGIBILITY:
Inclusion Criteria:

TRACERx Patients

* Multi-region sequencing data of the primary tumour available.
* TRACERx patients should be approached for a biopsy of the active locally advanced or metastatic disease but this is not mandated for DARWIN2 trial inclusion. Consent for this biopsy will be obtained within the TRACERx study.

Non-TRACERx patients

Minimum requirement:

• Fresh frozen biopsy of active locally advanced or metastatic disease OR at least two FFPE regions from primary tumour available

Optimal Tissue availability:

* Multi-region tissue of the primary tumour available (FFPE or fresh frozen) AND a fresh frozen biopsy of active locally advanced or metastatic disease
* OR One archival biopsy tissue sample (FFPE or fresh frozen)/pre-extracted DNA sample AND one fresh frozen biopsy of active locally advanced or metastatic disease
* OR Two fresh biopsies of active locally advanced or metastatic disease that are spatially separated e.g. one lymph node biopsy AND one lung biopsy.

Consent for the biopsy(ies) of the active locally advanced or metastatic disease for non-TRACERx patients must be taken using the DARWIN2 'trial entry tissue sample' consent form.

* Arm 1: Absence of any actionable mutation

  * ECOG PS 0-1 for MPDL3280A in combination with chemotherapy
  * ECOG PS 0-2 for MPDL3280A monotherapy.
  * Ability to avoid ibuprofen 2 days before, the day of, and 2 days following administration of Pemetrexed (combination therapy involving pemetrexed only)
  * Ability to take folic acid, Vitamin B12, and dexamethasone according to protocol (combination therapy involving pemetrexed only):
* Arm 2: Presence of BRAFV600 mutation

  - ECOG PS 0-2 for arm 2
* Arm 3: Presence of ALK/RET gene fusion and ALK IHC+/RET FISH

  - ECOG PS 0-2 for arm 3
* Arm 4: Presence of HER2 amplification and HER2 IHC 3+ only

  - ECOG PS 0-1 for arm 4.
* Absence of sensitising EGFR mutation (tested according to local protocol). The only exception will be patients who progress on DARWIN1 or on EGFR TKi off-study e.g. standard of care (if agreed following prior discussion with the CI & UCL CTC), or patients with squamous cell carcinoma
* Absence of ALK fusions (tested according to local protocol) except for patient being considered for arm 3. Patients with squamous cell carcinoma do not require local testing for EGFR sensitising mutations and ALK fusions prior to inclusion for the trial.
* Written Informed consent for DARWIN2.
* Measurable disease by RECIST v1.1. Patients without measurable disease may be eligible following discussion with the CI and UCL CTC but will not count towards the PFS primary endpoint. See Appendix 4.
* At least 18 years of age.
* Anticipated life expectancy of at least three months.
* Able to swallow and retain oral medication for arms 2 & 3.
* Adequate organ function as defined by the following baseline values:

  * Absolute neutrophil count (ANC) ≥1.5x109/L
  * Platelets ≥100x109/L
  * Serum bilirubin ≤1.5 x upper limit of normal (ULN). (In case of Gilberts syndrome discuss with TMG)
  * Aspartate aminotransferase (AST) or Alanine aminotransferase (ALT) ≤3xULN or ≤5x ULN if liver metastases are present). *
  * Creatinine clearance must be >30mL/min calculated or measured.
* Women with child-bearing potential, or men who are able to father a child, must be willing to practice highly effective methods of birth control during the trial and for 7 months after the end of treatment.
* Women of childbearing potential must have a negative pregnancy test within 14 days before registration.

Exclusion Criteria:

* Suitable for radical radiotherapy.
* Palliative radiotherapy within 1 week prior to registration.
* Patients with current or pre-existing interstitial lung disease.
* Patients with active pre-existing autoimmune disease (some exceptions allowed).
* Known hypersensitivity to study IMP or to any of the excipients
* Inability to understand or to comply with the requirements of the trial, trial protocol or to provide informed consent.
* Anti-cancer therapy including chemotherapy, radiation therapy (palliative dose within 7 days), immunotherapy (other than MPDL3280A (Atezolizumab) for Arm 1), biologic therapy, or major surgery within 14 days prior registration.
* Known human immunodeficiency virus (HIV), Hepatitis B Virus (HBV), Hepatitis C Virus (HCV) or syphilis infection. Subjects with evidence of hepatitis B virus clearance may be enrolled.
* History of other malignancy; Exception: (a) Subjects who have been successfully treated and are disease-free for 3 years, (b) a history of completely resected non-melanoma skin cancer, (c) successfully treated in situ carcinoma, (d) CLL in stable remission, or (e) indolent prostate cancer requiring no or only anti-hormonal therapy with histologically confirmed tumour lesions that can be clearly differentiated from lung cancer target and non-target lesions are eligible.
* Patients with symptomatic brain metastases.
* Severe symptomatic arrhythmias (excluding atrial fibrillation)
* The following cardiac abnormalities:

  * Corrected QT (QTc) interval ≥480 msecs (Arm 2)
  * Arm 4: LVEF <50%
  * History of acute coronary syndromes (including unstable angina) within the past 6 months
  * Coronary angioplasty, or stenting within the past 24 weeks
  * Class III, or IV heart failure as defined by the New York Heart Association (NYHA) functional classification system
  * History of known arrhythmias (except sinus arrhythmia and atrial fibrillation) within the past 3 months
  * History of myocardial infarction within the past 3 months
* Uncontrolled medical conditions (i.e., diabetes mellitus, hypertension, uncorrectable electrolyte abnormalities (including magnesium etc), psychological, familial, sociological, or geographical conditions that do not permit compliance with the protocol; or unwillingness or inability to follow the procedures required in the protocol.
* Pregnant, lactating or actively breastfeeding females.
* Arm 1: Treatment with systemic corticosteroids or other systemic immunosuppressive medications (including but not limited to prednisone, dexamethasone (>2mg), cyclophosphamide, azathioprine, methotrexate, thalidomide) within 2 weeks prior to registration, or anticipated requirement for systemic immunosuppressive medications during the trial

  * Patients who have received acute, low-dose, systemic immunosuppressant medications (e.g., a one-time dose of dexamethasone for nausea) may be enrolled in the trial after discussion with CTC.
  * The use of inhaled corticosteroids and mineralocorticoids (e.g., fludrocortisone) is allowed.
  * Low-dose supplemental corticosteroids for adrenocortical insufficiency are allowed. Doses of ≤2mg dexamethasone or equivalent (e.g. ≤12.5mg prednisolone) are allowed.
* Arm 1 (combination therapy involving pemetrexed only): Presence of third space fluid which cannot be controlled by drainage before or during initiation of pemetrexed therapy
* Arm 1 (combination therapy involving pemetrexed only):

  * Bilirubin >1.5 times the upper limit of normal
  * Transaminases >3.0 times the upper limit of normal (ULN), except in presence of known hepatic metastasis, wherein may be up to 5 times the ULN
* Arm 1: Patients cannot receive MPDL3280A (Atezolizumab) monotherapy if their immediate previous line of treatment has contained immunotherapy targeting PDL1 or PD1 with or without chemotherapy, see Appendix 6 (3).
* Arm 1: Patients cannot receive MPDL3280A (Atezolizumab) in combination with chemotherapy if their immediate previous line of treatment has contained immunotherapy targeting the PDL1 or PD1 given in combination with chemotherapy, see Appendix 6 (3).
* Arm 2: Previous BRAF inhibitor therapy.
* Arm 2: Patients taking medicines known to prolong QT interval 2 weeks prior to registration. Use also not permitted while on trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2017-05-12 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Progression free survival (PFS) | From date of registration until the date of first documented progression or death (whichever occurs first), assessed up to 84 months
  Defined as the period between the date of registration to the date of subsequent progression or death (whichever occurs first)
Overall survival | From date of registration until death date, assessed up to 84 months
  Time to event outcomes

SECONDARY OUTCOMES:
Objective response rate | From date of registration until last CT scan, assessed up to 84 months
  Investigator-assessed according to RECISTv1.1 and irRC (Arm 1 only)
Progression | From date registration until progression, , assessed up to 84 months
  ime to event outcomes
Duration of response | Period between first complete response or partial response until the first date recurrence or progressive disease, assessed up to 84 months
  Period between first complete response or partial response until the first date recurrence or progressive disease, assessed up to 84 months
Toxicity - Dose reductions, interruptions, modifications and exposure | From date of regsitration until end of treatment, assessed up to 84 months
  Dose reductions, interruptions, modifications and exposure
Exploratory assessments | Assessed at end of trial, at approximately 84 months
  Interrogation of recurrence and progression biopsies to decipher the molecular basis for resistance in combination with analyses of CTCs/cfDNA as well as CT imaging heterogeneity analyses

CONTACTS AND LOCATIONS:
Overall Officials: Charles Swanton, Principal Investigator — UCL
Locations (1):
- Univeristy College London Hospital, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No